CLINICAL TRIAL: NCT03072095
Title: Patient-Centered Outreach to Increase Colorectal Cancer Screening in a Community Health Setting
Brief Title: Colorectal Cancer Screening in a Community Health Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Shivan J Mehta, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 826576
Record Dates: First submitted 2017-02-23; First posted 2017-03-07 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Cancer of the Colon
Keywords: Colorectal Neoplasms; Colonic Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Rectal Diseases
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Rectal Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text-only (Experimental): Text-only outreach
  Interventions: Behavioral: Text-only
- Text + Lottery (Experimental): Text outreach + financial incentive
  Interventions: Behavioral: Text + Lottery

INTERVENTIONS:
Behavioral: Text-only — Subjects will receive a text communication indicating they are overdue for colon cancer screening with the option to elect to receive a free, at-home FIT kit.
  Arms: Text-only
Behavioral: Text + Lottery — Subjects will receive a text communication indicating they are overdue for colon cancer screening with the option to elect to receive a free, at-home FIT kit and a 1 in 5 chance to win a $100 gift card for completing the kit.
  Arms: Text + Lottery

SUMMARY:
This randomized controlled pilot study at the Health Annex, Family Practice & Counseling Network (FPCN), a community clinic in Southwest Philadelphia, aimed at providing data on the feasibility of a mailed FIT approach to CRC screening in a community health setting, and how patients respond to text messaging and behavioral economic engagement incentives.

DETAILED DESCRIPTION:
This is a single-center RCT at the Family Practice & Counseling Network (FPCN), a community clinic in Southwest Philadelphia with 320 eligible subjects between the ages of 50-74 randomized to two study arms:

1. text messaging outreach (text)
2. text messaging outreach with lottery for 1/5 chance to win a financial incentive (text + lottery).

Findings will provide data on the feasibility of this mailed FIT approach in a community health setting, and how patients respond to text messaging and behavioral economic engagement incentives.

ELIGIBILITY:
Inclusion Criteria:

1. Between 50 and 74 years old
2. Has active medical insurance
3. Has had had at least one visit at Health Annex in the prior 12 months (at time of chart review)
4. Due for CRC screening (no colonoscopy in last 10 years, sigmoidoscopy in last 5 years, or stool testing in last 1 year)
5. Asymptomatic for CRC

Exclusion Criteria:

1. Has had prior colonoscopy within 10 years, sigmoidoscopy within 5 years, and FOBT/FIT within twelve months of the chart review (we will exclude patients who self-report undergoing any of the above procedures)
2. Has a history of CRC
3. Has a history of other GI cancer
4. Has history of confirmed Inflammatory Bowel Disease (IBD) (e.g. Crohns disease, ulcerative colitis)
5. Has a history of colon polyps
6. Has had a colectomy
7. Has a first-degree relative that has been diagnosed with CRC
8. Has been diagnosed with Lynch Syndrome (i.e. HNPCC)
9. Has been diagnosed with Familial Adenomatous Polyposis (FAP).
10. Has iron deficiency anemia
11. Has recent history of lower GI bleeding
12. Has metastatic (Stage IV) blood or solid tumor cancer
13. Has end stage renal disease
14. Has had congestive heart failure
15. Has dementia
16. Has liver cirrhosis
17. Has any other condition that, in the opinion of the investigator, excludes the patient from participating in this study
18. Does not use a mobile phone enabled to send and receive text messages

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
FIT completion within 3 months | 3 months
  The percentage of participants who successfully complete the FIT

SECONDARY OUTCOMES:
Response to text-based CRC screening outreach | 3 months
  The percentage of people who respond to text message

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Family Practice & Counseling Network - Health Annex, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mehta SJ, Oyalowo A, Reitz C, Dean O, McAuliffe T, Asch DA, Doubeni CA. Text messaging and lottery incentive to improve colorectal cancer screening outreach at a community health center: A randomized controlled trial. Prev Med Rep. 2020 May 8;19:101114. doi: 10.1016/j.pmedr.2020.101114. eCollection 2020 Sep. PMID 32477853